CLINICAL TRIAL: NCT07195656
Title: Evaluation of a Non-Implanted Electrical Stimulation Device for Overactive Bladder (OAB) EVANESCE-II
Brief Title: Evaluation of a Non-Implanted Electrical Stimulation Device for Overactive Bladder (OAB)
Acronym: EVANESCE-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FemPulse Corporation (Industry)
Collaborators: Moxie Clinical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP012
Record Dates: First submitted 2025-09-24; First posted 2025-09-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Overactive Bladder (OAB)
Keywords: neuromodulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Device Group (Experimental): Subjects receiving the FemPulse System
  Interventions: Device: Device Group
- Medication Group (Other): Subjects receiving medication
  Interventions: Drug: Medication Group

INTERVENTIONS:
Device: Device Group — non-implanted, vaginal electrical stimulation device
  Arms: Device Group
Drug: Medication Group — OAB Medication
  Arms: Medication Group

SUMMARY:
A study to evaluate the safety and effectiveness of FemPulse System

ELIGIBILITY:
Key Inclusion Criteria:

* Females, defined as a person with a uterus and cervix, ≥21 years old, with a diagnosis of OAB and symptoms for more than 6 months, as confirmed by a physician. OAB is defined by urinary urgency, usually with urinary frequency and nocturia, with or without urgency urinary incontinence with symptoms
* Willing and able to comply with study required procedures and visits (e.g., maintaining consistent medication use, fluid intake, diary completion).

Key Exclusion Criteria:

* Systemic condition or disease that may interfere with study participation (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction, etc.) as determined by study investigator.
* Not an appropriate study candidate as determined by investigator.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 151 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Voids per Day | 6 months
  Difference in mean change between device and medication groups in number of voids per day (VPD)

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Sutherland, MD, Principal Investigator — FemPulse Corporation
Locations (15):
- United States (15):
  - Cedars Sinai, Beverly Hills, California
  - UCLA, Los Angeles, California
  - UC Irvine, Orange, California
  - Stanford, Palo Alto, California
  - USCD, San Diego, California
  - Holy Cross Medical Group - Women's Center, Fort Lauderdale, Florida
  - Comprehensive Urologic, Barrington, Illinois
  - University of Louisville, Louisville, Kentucky
  - Chesapeake Urology, Owings Mills, Maryland
  - Minnesota Urology, Woodbury, Minnesota
  - Adult & Pediatric Urology, Omaha, Nebraska
  - Atrium Health, Charlotte, North Carolina
  - Southern Urogynecology, West Columbia, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - INOVA, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No